CLINICAL TRIAL: NCT01011803
Title: Correlation of Phonation With Deglutition and Aspiration Risk in the ICU Patients - an Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Emir Festic, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 09-004079-05
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Aspiration
Keywords: Deglutition; Phonation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined speech therapy tools, measures of swallowing function (Experimental): All subjects will be assessed using combined speech therapy tools and ordinal measures of swallowing function. The combined speech therapy tools were [diadochokinesis, glottal coup, and the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V)]. The ordinal measures of swallowing function included Dysphagia Admission Screening Tool (DAST), Modified Barium Swallow (MBS), and Fiberoptic Endoscopic Evaluation of the Swallow (FEES).
  Interventions: Other: Combined speech therapy tools, measures of swallowing function

INTERVENTIONS:
Other: Combined speech therapy tools, measures of swallowing function — All subjects will be assessed using combined speech therapy tools and ordinal measures of swallowing function. The combined speech therapy tools were [diadochokinesis, glottal coup, and the Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V)]. The ordinal measures of swallowing function included Dysphagia Admission Screening Tool (DAST), Modified Barium Swallow (MBS), and Fiberoptic Endoscopic Evaluation of the Swallow (FEES).

SUMMARY:
Swallowing implies the appropriate use and sufficient function of specific muscles that are also used in speech. Theoretically, if these muscles are functionally affected then phonation and vocalization should be impaired, as well. The purpose of this study is to examine the relationship between functions of speech and risk of aspiration as defined by swallowing function, and to investigate the diagnostic potential that functions of speech may have in predicting the risk of aspiration. This could allow for earlier stratification of ICU patients for aspiration risks. Aspiration pneumonia has been reported in more than 20% of patients with health care-associated pneumonia. There are multiple tools to assess for risk of aspiration in the ICU, yet these are time consuming, often delayed and involve advanced testing that is performed by a certified speech-language pathologist and/or radiologist. A novel 3-step phonetic evaluation was created and will be implemented on ICU patients at risk for aspiration, and the results will be correlated to the standard swallowing tests. If strong correlation is found in this pilot study, then formal clinical trial will follow to confirm that the simple bed-side phonetic evaluation could allow for earlier identification of patients at risk for aspiration, and more efficient management relative to time and resources utilization.

DETAILED DESCRIPTION:
Aspiration is defined as entry of a solid or liquid material into the respiratory tract, below the vocal folds, or inhalation of fumes and vapors. Aspiration pneumonia is an infectious process caused by aspirated oropharyngeal flora, while aspiration pneumonitis is caused by a direct chemical insult due to the aspirated material.

Aspiration pneumonitis and pneumonia among hospitalized patients result in increased morbidity, mortality and utilization of resources, with increased costs of care. Early identification of patients at risk for aspiration is crucial to prevent this preventable and often iatrogenic condition.

In general, the most common predisposing factors for aspiration in adults are alcoholism, stroke, neuromuscular disorders, seizures, and loss of consciousness, and these patients are usually cared for in the ICU setting. Furthermore, critically ill patients are also at risk as they are frequently under varying degrees of sedation, especially early in the post extubation period. Postoperative patients in addition may have prolonged functional dysphagia due to lingering effect of neuromuscular blocking agents. However, risks of aspiration may apply to any hospitalized patient and further studies with broader inclusion criteria will be needed based on the preliminary results of this pilot study.

There are multiple tools to assess for risk of aspiration in the ICU. These include Dysphagia Admission Screening Tool (DAST), Fiberoptic Endoscopic Evaluation of the Swallow (FEES) and Modified Barium Swallow (MBS), which are routinely performed at our institution. The DAST is relatively novel screening tool, brought up as an early method for identification of dysphagia, as mandated by Joint Commission. This test has not been yet validated. It was created in 2004 in order to reduce the risk of aspiration among new stroke patients, based upon literature review, research and a strong foundation of knowledge and experience in Speech-Language Pathology in evaluating dysphagia. The FEES and MBS are time consuming, often delayed and involve advanced testing that is performed by a certified speech-language pathologist and/or radiologist. MBS also requires transport of the patient from the ICU to the radiology suite and back. These tests examine function of swallow mechanism in order to predict individual patient's risk of aspiration. They are reported as pass or fail and graded from 1-8, depending on the degree of the bolus penetration into the airway and/or expulsion from the airway. The current "gold standard" to determine the risk of aspiration is considered to be MBS.

We hypothesize that among critically ill, impairments in phonation correlate significantly to impairments in deglutition. Since in current practice patient's risk for aspiration is judged based on swallowing ability, strong correlation between impairments in speech and swallow mechanisms may allow prognostication based on phonation assessment alone. As the phonetic evaluation is simple, bedside test, it may result in earlier identification of the patient at risk for aspiration and obviate need for additional, invasive and expensive tests, and additional staff utilization for patient transport, testing and interpretation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients admitted to the ICU, deemed at risk for aspiration, who require FEES and MBS per speech therapy evaluation.
2. Ability to follow commands, read English language, vocalize and complete a predefined phonation test and the DAST.
3. Patients are able to undergo formal swallow evaluation by FEES and/or MBS.

Exclusion Criteria:

1. Patients who have had any type of head and neck surgery.
2. Patients that cannot read or talk, or speak/understand English language.
3. Patients with delirium, disorientation, unable to follow commands.
4. Patients with gastric tubes, tracheostomy or strict order for nothing by mouth.
5. Coagulation disorder that is prohibitive for FEES (platelets <50, 000, ongoing or uncontrolled bleeding, international normalized ratio (INR)> 1.5, activated partial thromboplastin time (aPTT) greater than 1.5 times normal value).
6. Patients that cannot sit up at 90 degrees for MBS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Ability of combined speech score to predict moderate to severe MBS/FEES Dysphagia | 24 hours
  Associations between measures of speech functions and ordinal measures of swallowing function will be examined by estimating Pearson's correlation coefficient. Categorical variables will be summarized with number and percentage.

SECONDARY OUTCOMES:
Ability of each individual speech score to predict MBS/FEES Dysphagia | 24 hours
  Associations between measures of speech functions and ordinal measures of swallowing function will be examined by estimating Pearson's correlation coefficient. Categorical variables will be summarized with number and percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Emir Festic, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States